CLINICAL TRIAL: NCT00044603
Title: Vulnerability of the Fetus/Infant to PAH, PM2.5 AND ETS
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 10165-CP-001
Record Dates: First submitted 2002-09-03; First posted 2002-09-05 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Pregnancy
Keywords: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biologic samples were collected from the mothers and their children as follows: maternal blood (30-35 ml) within 1 day postpartum and umbilical cord blood (30 - 60 ml) collected by delivery room staff immediately after the cord was cut. Members of the research staff transported the samples to the laboratory immediately. The buffy coat, packed red blood cells, and plasma samples were separated and stored at -70°C and then shipped to Columbia University. Placental tissue and meconium were also collected. The placental tissue and meconium were sent to Columbia and stored for future analysis under separate funding.
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to examine the effects of in utero and postnatal exposure to environmental pollutants in a cohort of pregnant women and their newborns in Krakow, Poland

DETAILED DESCRIPTION:
There is growing concern about adverse developmental effects in infants and young children from prenatal exposure to environmental air pollutants, including polycyclic aromatic hydrocarbons (PAH), particulate matter (PM2.5), and environmental tobacco smoke (ETS). The proposed study combines expertise in molecular epidemiology and biomarkers, state-of- the-art pollutant monitoring techniques, and a strong theoretical framework to guide assessment of the impacts of these pollutants on fetal and child growth and development. The specific aims are: 1. To test the hypothesis that prenatal exposure to airborne polycyclic aromatic hydrocarbons (PAH) adversely affects fetal growth and early childhood growth and development, after controlling for non-PAH components of PM2.5, ETS, nutritional status (essential fatty acids and antioxidants) and other potential confounders; 2. To explore whether non-PAH components of PM2.5, and ETS have an independent effect on birth outcomes and childhood growth and development, after controlling for PAH, and to explore possible interactions between PAH, PM2.5 and ETS; and 3. To estimate the relative contribution of ambient PAH pollution vs. ETS and other indoor PAH sources to a) personal PAH exposure and PAH-DNA adducts and b) impairment of fetal growth and early child development. To achieve these aims, the international team of researchers will carry out a prospective cohort study of 400 nonsmoking pregnant women living in Krakow, Poland, and will follow their newborns for 12 months postnatally. Fetal growth will be assessed at birth by weight, length, head circumference, and size for gestational age. Childhood growth and developmental outcomes will be measured using the Fagan Test and the Bayley Scales. Strengths of the research include the combination of personal inhalation monitoring of PAH and PM2.5 with biomarkers (umbilical cord blood levels of PAH-DNA adducts, cotinine, essential fatty acids, antioxidants and lead) to estimate in utero exposure to the pollutants of interest and potential confounders. The Polish cohort provides a valuable model for study since emissions from coal burning and traffic are relatively high. However, the results will be broadly applicable since exposures to PAH, ETS and PM2.5 during pregnancy are common in virtually all industrialized regions of the world. It is anticipated that this research will provide relevant data to policymakers concerned with protecting the health of young children.

ELIGIBILITY:
Inclusion criteria:

* Pregnant women between 18 and 40 years old
* Resided for at least 1 year within proximity to air monitoring station

Exclusion criteria:

* Smoking/ illicit drugs
* Hypertension
* Diabetes
* Occupational exposure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Only Polish and Caucasian women and their children are included in the study. There are no race/ethnic minorities included because the Krakow population is ethnically and racially homogeneous (almost 100% Caucasian).
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2000-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Fetal growth | Birth
  Fetal growth is assessed at birth by weight, length, head circumference, and size for gestational age

SECONDARY OUTCOMES:
Childhood growth and neurodevelopmental outcomes | 3 months - 3 years
  At 6 months of age, information regarding physical growth was collected from pediatric assessment and neurobehavioral development was evaluated using the Fagan Test of Infant Intelligence. At one year of age and annual time intervals thereafter, physical growth was assessed during a pediatric examination and neurobehavioral development was assessed with the Bayley Scales of Infant Development.

CONTACTS AND LOCATIONS:
Overall Officials: Frederica P Perera, DrPH, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, 722 W 168th St, 12th Floor, New York, New York, United States